CLINICAL TRIAL: NCT01955772
Title: Randomized, Prospective, Multicenter Study to Compare Enteral Nutrition to Parenteral Nutrition as Feeding Support in Patients Presenting Malignant Hemopathy Who Underwent an Allogeneic Hematopoietic Stem Cell Transplantation.
Acronym: NEPHA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Societe Francaise de Greffe de Moelle et de Therapie Cellulaire (Other); Société Francophone Nutrition Clinique et Métabolisme (Other); Laboratoires NUTRICIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0165; 2011-A1288-33
Record Dates: First submitted 2013-07-19; First posted 2013-10-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Myeloablative Allo-SCT
Keywords: Haematopoietic stem cell transplantation; Malignant hemopathy; Artificial nutrition
MeSH Terms: interventions — alanylglutamine

ARMS (2):
- EN (Enteral Nutrition) (Experimental): NE group: According to the HAS and SFNEP recommendations and the good practice rules, a polyurethane or silicone NGT, 8 to 10 French units, will be inserted and its positioning will be controlled by radiography before the EN beginning. Polyurethane and silicone are very well tolerated by nasal and oesophagus mucosa and have a long life duration allowing keeping the same tube during 2 to 3 months.
  PN group: PN will be administrated by a central venous catheter, which is usually inserted in allo-HSCT patients to allow the administration of chemotherapy and of the different parenteral treatments.
  Interventions: Drug: Enteral nutrition alanyl-glutamin, Dipeptiven
- PN (Parenteral Nutrition) (Other): NE group: According to the HAS and SFNEP recommendations and the good practice rules, a polyurethane or silicone NGT, 8 to 10 French units, will be inserted and its positioning will be controlled by radiography before the EN beginning. Polyurethane and silicone are very well tolerated by nasal and oesophagus mucosa and have a long life duration allowing keeping the same tube during 2 to 3 months.
  PN group: PN will be administrated by a central venous catheter, which is usually inserted in allo-HSCT patients to allow the administration of chemotherapy and of the different parenteral treatments.
  Interventions: Drug: Enteral nutrition alanyl-glutamin, Dipeptiven

INTERVENTIONS:
Drug: Enteral nutrition alanyl-glutamin, Dipeptiven — Enteral nutrition versus parenteral nutrition
  Other Names: All patients will received, whatever treatment arm, intravenous alanyl-glutamin, Dipeptiven which have AMM.

SUMMARY:
Myeloablative allogeneic hematopoetic stem cell transplantation (AHSCT) are prone to frequent secondary malnutrition to metabolic and digestive troubles due to conditioning regimen, treatments (antibiotics, immunosuppressive therapy…) and graft complications (graft versus host disease). In the absence of appropriate nutritional support, myeloablative conditioning lead to a rapid serious denutrition. But, it is known as negative independent prognostic factor of overall survival of patients who presented malignant hemopathy treated by high-dose chemotherapy or AHSCT. Furthermore, it increases hospitalisation delay and decreases quality of life. In AHSCT with myeloablative conditioning, introduction of nutritional support is recommended. However, type of nutritional support remains not clearly defined. Parenteral nutrition is user but favour infections and secondary effects potentially decrease by intravenous glutamine. Few previous studies with low number of patients, mainly retrospective or combining allo-and auto HSCT had shown feasibility, acceptable tolerance and low cost of enteral nutrition (EN). A recent prospective no-randomized study in 45 adults patients who had undergone AHSCT with myeloablative conditioning find a significant decrease of day-100 mortality (5% vs 30%), of infection mortality, of median duration of parenteral nutrition (PN) and prevalence of GvH (Graft versus Host Disease) grade III-IV in EN (enteral nutrition) group. These results had to be confirmed by a randomized study. As EN is 4 to 5 more cheaply than PN, besides mortality/morbidity stakes for the patient, this study could have potential economic interest.

DETAILED DESCRIPTION:
EN (enteral nutrition) or PN (parenteral nutrition) artificial nutrition will be launched at D1-D2 of the transplantation (D0 being the day of the transplantation),without taking into account the oral intake. This helps in particular to launch the EN after the stage of significant digestive problems related to the conditioning and before the mucositis appearance.

EN group: According to the HAS and SFNEP (Societe francophone nutrition clinique) recommendations and the good practice rules, a polyurethane or silicone NGT(Naso gastric tube), 8 to 10 French units, will be inserted and its positioning will be controlled by radiography before the EN beginning. Polyurethane and silicone are very well tolerated by nasal and oesophagus mucosa and have a long life duration allowing keeping the same tube during 2 to 3 months.

PN group: PN will be administrated by a central venous catheter, which is usually inserted in allo-HSCT patients to allow the administration of chemotherapy and of the different parenteral treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Men and women
* Patients undergoing myeloablative allo-SCT
* Allo-SCT genoidentical or phenoidentical 10/10
* Patients affiliated with a social security organisation
* Patients having signed the informed consent

Exclusion Criteria:

* Status of tumour progression at the moment of the allo-SCT
* Artificial nutrition begun before the inclusion
* Inability to understand the protocol (linguistic barrier, cognitive difficulties)
* Contraindication or associated pathology that does not allow to carry out EN or PN according to the protocol
* Medical history of progressive psychiatric illness
* Medical history of another progressive cancer or occurrence in the 5 previous years
* Presence of a simultaneous serious and uncontrolled disease such as severe cardiac, renal, hepatic or respiratory failure or severe sepsis
* Previous allo-SCT
* Participation in another clinical trial studying an allograft procedure, and applying modalities that are not available in routine practice (including innovative immunosuppression and graft or conditioning regimens not considered as myeloablative)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Mortality related to the transplant | at day 100

SECONDARY OUTCOMES:
Occurrence of post-transplant complications targeting acute GVH, mucite and infections | 12 months after AHSCT (hematopoietic stem cell transplantation)
Overall survival and disease free survival | 12 months after AHSCT (hematopoietic stem cell transplantation)
Evolution of nutritional state | 12 months after AHSCT
  All patients will received, whatever treatment arm, intravenous alanyl-glutamin, Dipeptiven which have AMM.
Tolerance of nutritional support mainly on digestive and hepatobiliary disorders | 12 months after AHSCT
  All patients will received, whatever treatment arm, intravenous alanyl-glutamin, Dipeptiven which have AMM.
Engraftment rates | Day30, Day60, Day90 and Day180
quality of life assessment | Day7, Day90, Day180 and Day360

CONTACTS AND LOCATIONS:
Overall Officials: Corinne BOUTELOUP, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Lemal R, Cabrespine A, Pereira B, Combal C, Ravinet A, Hermet E, Bay JO, Bouteloup C. Could enteral nutrition improve the outcome of patients with haematological malignancies undergoing allogeneic haematopoietic stem cell transplantation? A study protocol for a randomized controlled trial (the NEPHA study). Trials. 2015 Apr 7;16:136. doi: 10.1186/s13063-015-0663-8. PMID 25872934